CLINICAL TRIAL: NCT05575804
Title: Phase Ib/II Study of GQ1001 and Pyrotinib in HER2 Positive Metastatic Breast Cancer Patients Who Had Failed Previous Anti-HER2 Treatment（GRACE）
Brief Title: GQ1001 Combined With Pyrotinib for Treatment With HER2 Positive Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: GeneQuantum Healthcare (Suzhou) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRACE
Record Dates: First submitted 2022-10-05; First posted 2022-10-12 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Advanced/ Metastatic Her-2 Positive Breast Cancer
Keywords: HER2-ADC; pyrotinib; Advanced/ Metastatic Her-2 positive Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients will receive the recommended phase 2 dose of GQ1001 determined in phase I. GQ1001 infusions on day 1 of each 21-day cycle combinate with pyrotinib 320mg orally once daily until disease progression or unacceptable toxicity.
  Interventions: Drug: GQ1001+pyrotinib
- control group (Active Comparator): Patients will receive pyrotinib 400mg orally once daily in combination with capecitabine 1000mg/m2 twice daily, day1-14, every three weeks until disease progression or unacceptable toxicity.
  Interventions: Drug: pyrotinib+capecitabine

INTERVENTIONS:
Drug: GQ1001+pyrotinib — GQ1001 infusions on day 1 of each 21-day cycle combinate with pyrotinib 320mg orally once daily until disease progression or unacceptable toxicity. I.
  Arms: experimental group
Drug: pyrotinib+capecitabine — pyrotinib 400mg orally once daily in combination with capecitabine 1000mg/m2 twice daily, day1-14, every three weeks until disease progression or unacceptable toxicity.
  Arms: control group

SUMMARY:
The aim of this trial is to study the safety, pharmacokinetics and preliminary efficacy of the HER2-targeted antibody-drug conjugate GQ1001 in combination with pyrotinib in patients with HER2-positive metastatic breast cancer patients who had failed previous anti-HER2 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to provide written informed consent.
2. Men or women aged 18-75.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy greater than 3 months.
5. Left ventricular ejection fraction (LVEF) ≥50%.
6. Histopathological and/or cytological confirmed Her2-positive locally advanced or metastatic breast cancer (IHC3+, or IHC2+ and ISH+)
7. Failure for at least 1 line of standard systemic treatment for metastatic disease. Meet one of the following conditions:

1) Recurrent within 12 months after completing or during neoadjuvant/ adjuvant therapy (the regimens contain trastuzumab or its biosimilar with pertuzumab or not).

2) Received at least one treatment with trastuzumab or its biosimilar ±pertuzumab (monotherapy or in combination with other drugs) for recurrent or metastatic disease.

8. Previous exposure to taxanes. 9. Having at least one measurable lesion according to RECIST 1.1 . 10. Having sufficient bone marrow, liver and kidney functions: white blood cell count≥ 3×109/L; Absolute neutrophil count ≥ 1.5×109/L; Platelet count ≥ 100×109/L; Hemoglobin ≥ 9.0 g/dL with no blood transfusion in the past 28 days; Total bilirubin ≤ 1.5 x the upper limit of normal (ULN); AST and ALT ≤ 3.0 x ULN (or ≤ 5.0 x ULN in the presence of liver metastases); Serum creatinine ≤1.5 x ULN; Coagulation function (prothrombin time and activated partial thromboplastin time ≤1.5 x ULN); 11. Adequate wash-out periods: Major surgery ≥4 weeks; radiotherapy ≥4 weeks; targeted therapy or chemotherapy≥4 weeks; endocrine therapy≥2 weeks; targeted therapy and endocrine therapy≥2 weeks; mAbs and immunotherapy ≥4 weeks; Any investigational agents≥4 weeks; potent CYP3A4 inhibitor≥3*t1/2 weeks.

12. Female subjects must meet the following conditions: infertility or fertility and use high-efficiency contraceptive measures during the study and for 6 months following the last dose of the study drug infusion.

Exclusion Criteria:

1. Have active brain parenchymal metastasis. Patients with clinically stable brain parenchymal metastases can be included, including asymptomatic brain metastases that have not received local treatment; or patients who have previously received central nervous system metastasis therapy (radiotherapy or surgery), if imaging confirms that stability has been maintained for at least 4 weeks, and have stopped symptomatic treatment (including hormones and mannitol, etc.) for more than 4 weeks CNS (central nervous system) metastasis with clinical symptoms;
2. Have previously been treated with: another antibody-drug conjugate (ADC) consisting of DM1 or its derivative; previously received capecitabine (end of adjuvant therapy>1 year and not receive capecitabine after relapse were allowed); previously received pyrotinib (end of (neo)adjuvant therapy>6 months and no pyrotinib treatment after relapsed were allowed; received pyrotinib in metastatic settings and stopped for reasons other than disease progression and had disease progression after 6 months were allowed.
3. Have other malignant tumors within 5 years before signing the informed consent form ( except for cured skin basal cell carcinoma and cervical carcinoma in situ).;
4. The toxicity of previous anti-cancer therapy has not recovered to ≤1 as specified in CTCAE v5.0 (except for hair loss); chronic grade 2 toxicity might be determined per the investigator's judgment.
5. History of allergic reaction to any component of GQ1001.
6. Have a medical history of myocardial infarction, symptomatic congestive heart failure (CHF) (NYHA classes II-IV), unstable angina or serious cardiac arrhythmia within 6 months.
7. Have a corrected QT interval (QTc) prolongation to > 450 milliseconds (ms) in males and > 470 ms in females.
8. Have a history of (noninfectious) interstitial lung disease (ILD)/pneumonitis requiring steroids, current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
9. The cumulative dose of anthracyclines or equivalent>500 mg/m2.
10. Active and clinically significant bacterial, fungal or viral infection including hepatitis B (HBV), and hepatitis C (HCV).
11. Pregnancy or lactation.
12. Male or female subjects unwilling to use approved contraceptive methods (e.g. birth control pills, barrier device, intrauterine device, abstinence) during the study and for 7 months following the last dose of the study drug infusion.
13. Other circumstances that are deemed not appropriate for the study.
14. Inability to swallow, chronic diarrhea and intestinal obstruction, or other factors that affect drug administration and absorption.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs), Phase I | From the first dose to the end of Cycle 1, 21 days
  Side effects of drug or treatment that are serious enough to prevent an increase in dose or level of that treatment, according to NCI-CTCAE Version 5.0.
Maximum Tolerated Dose (MTD), Phase I | From the first dose to the end of Cycle 1, 21 days
  Highest administered dose with < 33% of participants experiencing dose-limiting toxicity (DLT) in the first 6 DLT evaluable participants.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 24 months
  Incidence and severity of Treatment-emergent adverse events, treatment-related adverse events and serious adverse events, according to NCI-CTCAE Version 5.0 (The number of participants who had treatment-related side effects in the population who had received one therapy at least).
Objective Response Rate (ORR), Confirmed by the researcher's evaluation, Phase II | up to 24 months
  The objective response rate will be analyzed according to the RECIST 1.1 standard tumor evaluation.

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax), Phase I | At the end of Cycle 3 (each cycle is 21 days)
  Maximum Serum Concentration (Cmax) of GQ1001, DM1, pyrotinib, and total anti-HER2 antibody
Trough Serum concentration (Cthough), Phase I | At the end of Cycle 3 (each cycle is 21 days)
  Trough Serum concentration (Cthough) of GQ1001, DM1, pyrotinib, and total anti-HER2 antibody
Area Under the Concentration-time Curve (AUC), Phase I | At the end of Cycle 3 (each cycle is 21 days)
  Area Under the Concentration-time Curve (AUC) of GQ1001, DM1, pyrotinib, and total anti-HER2 antibody
Objective Response Rate (ORR), Phase I | up to 24 months
  The objective response rate will be analyzed according to the RECIST 1.1 standard tumor evaluation.
Duration of Response (DoR) | up to 24 months
  DOR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death.
Disease Control Rate (DCR) | up to 24 months
  DCR is defined as the rate of the sum of CR, PR and SD according to the RECIST 1.1 standard tumor evaluation.
PFS | up to 24 months
  Progression-free survival (PFS) refers to the time from the date of randomization to the first researcher's evaluation of disease progression or death (calculated by the event that occurred first). The disease progression will be evaluated by the researchers according to the RECIST 1.1 standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China